CLINICAL TRIAL: NCT07204808
Title: A Comparative Study of High Velocity Resistance Training Versus Otago Exercise Training on Falling Risk in Elderly : A Randomized Controlled Trial
Brief Title: High Velocity Resistance Training Versus Otago Exercise Training on Falling Risk in Elderly
Acronym: HVRT/OTAGO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Shaimaa abu bakr bakr taha, Demonstrator, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Falling risk
Record Dates: First submitted 2025-09-23; First posted 2025-10-02 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Falling Risk

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago group (Active Comparator): Participants who will be randomized to the otago exercise program will receive an exercise program that include 17 exercises 5 for strengthen , 12 balance exercise and will starting and ending with a 2-to 3-min warm-up/cool-down period OEP consists of strengthening and balance exercises. Strengthening of ankle plantar and dorsiflexors, knee extensors and flexors, and hip abductors will be focused in traises. The progression will be performed by increasing the duration and then weights. Stair walking, sit-to-stand, heel-to-toe walking backward, toe walking, heel walking, one-leg stands, tandem walking, tandem stance, sideways walking, turning around, walking backward, walking, and knee bends were used for balance exercises. Three levels will be used for balance exercises: Level 1 will be 2 hands holding on, Level 2 will be one hand holding on, and Level 3 will be no hands or support. The individuals will repeat exercise 10 times session twice a week over 8 weeks
  Interventions: Device: High velocity resistance training + Otago Exercise Program
- High velocity resistance training group (Active Comparator): Participants who will be randomized to the HVRT will receive an exercise program targeting the lower limbs, to be performed twice a week for 8 weeks. Participants will be instructed to perform the exercises in a rapid and explosive manner such that all repetitions for each shortening phase (concentric activation of the muscle) will be performed as quickly as possible while the lengthening phase of the muscle (eccentric phase) will be controlled over 2-3 s
  Interventions: Device: High velocity resistance training + Otago Exercise Program

INTERVENTIONS:
Device: High velocity resistance training + Otago Exercise Program — Participants who will be randomized to the HVRT will receive an exercise program targeting the lower limbs, to be performed twice a week for 8 weeks. Participants will be instructed to perform the exercises in a rapid and explosive manner such that all repetitions for each shortening phase will be performed as quickly as possible while the lengthening phase of the muscle will be controlled over 2-3 s The exercise will be done (bilateral leg press, step up, sit to stand, calf raise). The 8 weeks will be divided in three phases .
  OEP consists of strengthening and balance exercises. Strengthening of ankle plantar and dorsiflexors, knee extensors and flexors, and hip abductors will be focused in this program. Ankle weight cuffs (1-3 kg) provide resistance for hip and knee exercises. The ankle plantar and dorsiflexors will be strengthened by performing heel and toe raise .
  plantar and dorsiflexors will be strengthened by performing heel and toe

SUMMARY:
The study aim is to find out the difference between applying the otago exercise training versus high velocity resisted training on risk of fall in elderly. There will be no significant difference between the effect of otago exercise program versus high velocity resisted training on risk of fall in elderly . 40 Old aged persons of both sex their age >65 years and have risk of falling will be recruited in this study.

DETAILED DESCRIPTION:
Type of study : Randomized trail This prospective interventional study that will be conducted on 40 case of both sex their age above 65

They randomly assigned into 2 equal groups:

Study group (A) 20 patients will receive otago exercise program and will do their normal activity of daily living. Study group (B) 20 patients will receive high velocity resisted training and will do their normal activity of daily living

ELIGIBILITY:
Inclusion Criteria:

* Age >65 years old.
* Both sex.
* Have limited their activity level due to concern about falling (with or without falling) score by short -FES > 7 and by
* fall risk check list ≥ 4.
* Participants will be independently ambulating

Exclusion Criteria:

* Any uncontrolled non musculoskeletal conditions that would make testing difficult and uncomfortable such as chronic obstructive airways disease and/or congestive heart failure.
* A pre-existing neurological condition that affects lower-limb strength, balance and or ambulation (e.g., polio, stroke).
* Any uncontrolled musculoskeletal or orthopedic conditions that may affect ambulation (e.g. rheumatoid arthritis).
* Severe cerebrovascular or peripheral venous insufficiency.
* History of surgery within the past 6 weeks.
* Sensory impairments (vision, hearing, etc.) that affect communication
* Previous diagnosis of dementia.
* Hypotension (systolic blood pressure <90 mmHg, diastolic blood pressure <60 mmHg

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Berg balance scale | "Baseline (pre-intervention) and after 8 weeks of intervention"
  The scale will evaluate an individual's ability to maintain their balance while performing functional activities. It includes 14 items and each section is scored between 0 (worst) and 4 (best), and measures level of dependence/independence in positions such as standing from sitting, standing with feet together, standing in full balance position, balancing on one leg, as well as ability to change positions. High BBS score will indicate good balance. Participants will be classified based on BBS score as high fall risk, balance disorder (0-20 points), moderate fall risk, acceptable balance (21-40 points), and low fall risk, good balance (41-56 points)
Time up and go test | "Baseline (pre-intervention) and after 8 weeks of intervention"
  Timed Up and Go is a commonly applied screening tool that helps to identify patients that are likely to fall. The test will be conducted with the following rules: at first, the tested person will sit on a chair with their back on the backrest; then, on the command "START," they will get up and walk 3m (on a level floor at a normal pace); next, having crossed a line, they will take a 180-degree turn and will come back to the chair to sit down again. The time will be measured by a stopwatch when the patient is instructed on how the test should be done . A test result less than 10 sec indicate low risk of fall , 10-19 sec -a moderate risk of fall and more than 19 -ahigh risk of fall

SECONDARY OUTCOMES:
30 sec chair stand test | "Baseline (pre-intervention) and after 8 weeks of intervention"
Short fall efficacy scale | "Baseline (pre-intervention) and after 8 weeks of intervention"
6 mwt | "Baseline (pre-intervention) and after 8 weeks of intervention"
Fall Risk check list | "Baseline (pre-intervention) and after 8 weeks of intervention"
Four stage balance test | "Baseline (pre-intervention) and after 8 weeks of intervention"

CONTACTS AND LOCATIONS:
Overall Officials: Tamer Ibrahim Abo Elyazed, Professor, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-suef University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No